CLINICAL TRIAL: NCT02866136
Title: Conservative Treatments of Retinoblastoma
Acronym: RETINO2011
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Fondation Rothschild Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2011-05
Record Dates: First submitted 2016-07-27; First posted 2016-08-15 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Retinoblastoma; Children; Retinal Neoplasm
MeSH Terms: conditions — Retinoblastoma; Retinal Neoplasms | interventions — Etoposide; Carboplatin; Drug Therapy; Melphalan; Vincristine; Platinum Compounds; Lasers; Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- (IV)Intravenous chemotherapy, laser diode (Other): Group 1 - Multicentric non randomised, phase II study for patients with retinoblastoma (unilateral group A,B according to age, group C according to the age and the vitreous seeding or bilateral groups A,B and C excluding the bilateral groups D or patients with bilateral macular threat).
  Treatment by chemoreduction (VP16, carboplatin) followed by Carboplatin + laser day 1 (chemothermotherapy) without laser treatment at day 8 (decreasing laser sessions) combined to local treatments from third course (laser, cryoapplication, I125 radioactive plaques or intravitreal Melphalan).
  Interventions: Drug: VP16, carboplatin; Drug: Carboplatin + laser day 1 (chemothermotherapy); Device: Laser (local treatment); Device: cryoapplication (local treatment); Radiation: I125 radioactive plaques (local treatment); Drug: intravitreal Melphalan (local treatment)
- (IA) Intraarterial Melphalan (Other): Group 2 - Multicentric non randomised, phase II study for the patients with bilateral very asymmetric disease (group D retinoblastoma on one of the eye, and the other amenable to a local treatment without chemotherapy) or unilateral presentation group D and groups B/C according to the age and vitreous seeding.
  Treatment by Melphalan chemotherapy administered by superselective catheterization of the ophthalmic artery and combined to local treatments (laser, cryoapplication, I125 radioactive plaques or intravitreal Melphalan).
  Interventions: Drug: Melphalan; Device: Laser (local treatment); Device: cryoapplication (local treatment); Radiation: I125 radioactive plaques (local treatment); Drug: intravitreal Melphalan (local treatment)
- (IV-PM) Intravenous 3 drugs chemotherapy (Other): Group 3 - Multicentric non randomised, phase II study for the patients with bilateral group D retinoblastoma or with a group D retinoblastoma on the only remaining eye. Treatment by 6 cycles of three drugs (VP16, carboplatin, vincristin) regimen combined to local treatments from the third cycle (laser, cryoapplication, I125 radioactive plaques or intravitreal Melphalan).
  Interventions: Drug: VP16, carboplatin, vincristin; Device: Laser (local treatment); Device: cryoapplication (local treatment); Radiation: I125 radioactive plaques (local treatment); Drug: intravitreal Melphalan (local treatment)

INTERVENTIONS:
Drug: VP16, carboplatin — Systemic treatment : Intravenous injections, 2 cycles (21 days)
  Other Names: etoposide, vepesid, chemotherapy
  Arms: (IV)Intravenous chemotherapy, laser diode
Drug: Melphalan — intraarterial injections, 3 to 6 cycles (1 month)
  Other Names: Alkeran, chemotherapy
  Arms: (IA) Intraarterial Melphalan
Drug: VP16, carboplatin, vincristin — Systemic treatment : Intravenous injections, 6 cycles (21 days)
  Other Names: etoposide, vepesid, leurocristine, Oncovin, chemotherapy
  Arms: (IV-PM) Intravenous 3 drugs chemotherapy
Drug: Carboplatin + laser day 1 (chemothermotherapy) — Chemothermotherapy : Intravenous injection by carboplatin and Laser at day 1
  Other Names: Carbo-laser, platinum-based chemotherapy
  Arms: (IV)Intravenous chemotherapy, laser diode
Device: Laser (local treatment)
  Other Names: Laser diode
Device: cryoapplication (local treatment)
Radiation: I125 radioactive plaques (local treatment)
Drug: intravitreal Melphalan (local treatment)

SUMMARY:
Conservative treatments of retinoblastoma (RETINO 2011)

1. -Multicentric non randomised, phase II study for the patients treated by chemoreduction (VP16, carboplatin) followed by chemothermotherapy without laser treatment at day 8
2. -Multicentric non randomised, phase II study for the patients with bilateral very asymmetric dis-ease (Group D eye on one of the eye) or unilateral presentation groups B/C/D according to the age and vitreous seeding
3. - Multicentric non randomised, phase II study for the patients treated by 6 cycles of three drugs regimen and local treatments for bilateral group D eyes or on the only eye.

ELIGIBILITY:
Inclusion Criteria:

Study 1 inclusion criteria:

* Patients affected by unilateral retinoblastoma groups A, B (according to the age), group C (according to the age and vitreous seeding),or bilateral retinoblastoma groups A, B, C (excluding the eyes with macular threat and bilateral group D eyes or on the only remaining eye) amenable to a conservative treatment (at least on one eye in bilateral disease) but needing initial chemotherapy because of the location, the size of the lesion (more than 4 mm of diameter), a vision threat or risks of intravitreal relapse making those patients not amenable to chemothermotherapy first line.
* Patients less than six months of age with unilateral retinoblastoma groups B, C, D, or bilateral very asymmetric with one eye group D and the other amenable to local treatments without chemotherapy.
* Children from 0 to 6 years old.

Study 2 inclusion criteria:

* Patients affected by unilateral or bilateral retinoblastoma group B (according to the age), group C (according to the age and vitreous seeding), or group D.
* Patients affected by bilateral retinoblastoma very asymmetric with a group D eye that can be treated by intraarterial chemotherapy by Melphalan and the other amenable to local treatments without chemotherapy.
* Children from 6 months to 6 years old.

Study 3 inclusion criteria:

* Children affected of bilateral group D retinoblastoma or on the only eye amenable to conservative treatment.
* Children from 0 to 6 years old.

Common inclusion criteria:

* Patients not previously treated by chemotherapy or radiotherapy for this tumour or another cancer.
* No contra-indications to the study treatments
* Possible long term follow-up.
* Written informed consent of the parents or the legal representative.
* Patients having social security cover.

Exclusion Criteria:

Study 1 exclusion criteria:

* Patients for whom a local treatment is possible without initial chemotherapy (tumour smaller than 4 mm and located far from optic nerve head or macula).
* Patients with an unilateral group D with massive tumour or group E eyes needing enucleation first line or after initial chemotherapy (in case of buphthalmia or suspected optic nerve invasion or extrascleral extension).
* Patients affected by bilateral retinoblastoma very asymmetric with a group D eye that can be treated by intraarterial chemotherapy by Melphalan and the other amenable to local treatments without chemotherapy.
* Patients with bilateral retinoblastoma and bilateral group D eyes or on the only remaining eye or presenting a bilateral macular threat requiring conservative treatment by a 6 cycles, three drugs regimen.

Study 2 exclusion criteria:

* Patients with a unilateral group D (extensive) or B or C but covering the optic nerve head or group E eyes for which enucleation is warranted first line or after chemotherapy (in case of buphthalmia or suspected optic nerve invasion or extrascleral extension).
* Patients with unilateral group D eye with tumour volume of more than 50% of eye volume, for whom a massive choroidal invasion could be associated (on clinical or imaging criteria) and for which enucleation is warranted.

Study 3 exclusion criteria:

* Patients for whom a local treatment is possible without chemoreduction (tumour smaller than 4 mm, distant from macula and from optic nerve head).
* Patients affected by bilateral retinoblastoma very asymmetric with a group D eye that can be treated by intraarterial chemotherapy by Melphalan and the other amenable to local treatments without chemotherapy.
* Patients with bilateral retinoblastoma without macular threat or groups A, B, C than can be treated with chemoreduction by VP16 and Carboplatin then chemothermotherapy without laser at day 8.

Common exclusion criteria:

* Patients older than 6 years old.
* Patients with extraocular retinoblastoma.
* Patients with a disease being a contra-indication to chemotherapy.
* Patients anteriorly treated by chemotherapy.
* Patients anteriorly treated by external beam irradiation.
* Patients anteriorly treated for another cancer.
* Follow-up not possible due to geographic distance from the center or for social or psychological reasons.
* Parents not having accepted the therapeutic strategy after explanations by the investigator.
* Contra-indication to the use of one of the drugs used in the study.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Rate of enucleation and external beam irradiation | From first day of treatment to 18 months after the end of treatments

SECONDARY OUTCOMES:
Number of relapses diagnosticated by fundus examination under general anesthesia until the age of 4 years, and without general anesthesia for older patients | 5 years
  Number of fundus examination positives without clinical symptoms and number of patients treated after fundus examination-related treatment with a controlled disease.
Prospective evaluation of the systemic, ocular and general sides effects (short term) of the intravenous chemotherapy, intraarterial chemotherapy, combined to the local treatments as well as the intravitreal injections of Melphalan | 5 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 and types of adverse events occuring in order to reassess the benefice-risk scale (by Independent Data Monitoring Committee), for each arm of the study and for the whole study.
Prospective evaluation of the systemic, ocular and general sides effects (medium and long term) of the intravenous chemotherapy, intraarterial chemotherapy, combined to the local treatments as well as the intravitreal injections of Melphalan | 5 years
  Rate of patient with a progression disease and/or presenting a medium/long term adverse event(s) or a second cancer.
Response to intravitreal chemotherapy by Melphalan | 18 months
  Number of patients with uncontrolled disease (progression) and/or presenting Adverse Event(s) as assessed by CTCAE v4.0, related to intravitreal chemotherapy by Melphalan.
Radiation doses received during intraarterial procedures | 18 months
  Time of scopies during ophthalmic arterial catheterism, doses delivered by the machine, doses received on skin.
Number of patients presenting a long term second tumour | until 20 years old

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Aerts, MD, Study Director — Institut Curie - Paris - France; Catherine Devoldere, MD, Principal Investigator — Amiens (FR), University College Hospital; Isabelle Pellier, MD, Principal Investigator — Angers (FR), University College Hospital; Véronique Laithier, MD, Principal Investigator — Besançon (FR), Jean Minjoz Hospital; Celine De Bouyn-Icher, MD, Principal Investigator — Bordeaux (FR), Pellegrin Regional Hospital; Liana-Stephania Carausau, MD, Principal Investigator — Brest (FR), University College Hospital; Damien BODET, MD, Principal Investigator — Caen (FR), University College Hospital; Justyna Kanold, MD, Principal Investigator — Clermont-Ferrand (FR), University College Hospital; Claire Briandet, MD, Principal Investigator — Dijon (FR), Bocage University College Hospital; Dominique Plantaz, Prof., Principal Investigator — Grenoble (FR), University College Hospital; Hélène Sudour-Bonnange, MD, Principal Investigator — Lille (FR), Oscar Lambret Center; Christophe Piguet, MD, Principal Investigator — Limoges (FR), University College Hospital; Cécile Faure Conter, MD, Principal Investigator — Lyon (FR), Leon Berard Center; Carole Coze, MD, Principal Investigator — Marseille (FR), La Timone Children Hospital; Nicolas Sirvent, MD, Principal Investigator — Montpellier (FR), Arnaud de Villeneuve Hospital; Ludovic Mansuy, MD, Principal Investigator — Nancy (FR), University College Hospital; Estelle Thebaud, MD, Principal Investigator — Nantes (FR), University College Hospital; Marilyne Dupuy-Poiree, MD, Principal Investigator — Nice (FR), University College Hospital; Frederic Millot, MD, Principal Investigator — Poitiers (FR), University College Hospital; Claire Pluchart, MD, Principal Investigator — Reims (FR), Regional University College Hospital; chloé Puiseux, MD, Principal Investigator — Rennes (FR), University College Hospital; Pascale Schneider, Prof., Principal Investigator — Rouen (FR), University College Hospital; Jean-Louis Stephan, Prof., Principal Investigator — Saint-Etienne (FR), University College Hospital; Natacha Entz-Werle, MD, Principal Investigator — Strasbourg (FR), University College Hospital; Anne-Isabelle Bertozzi-Salamon, MD, Principal Investigator — Toulouse (FR), Children Hospital; Pascale BLOUIN, MD, Principal Investigator — Tours (FR), University College Hospital; Michel Piotin, MD, Principal Investigator — Paris (FR), Adolphe Rothschild Ophtalmologic Foundation
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).